CLINICAL TRIAL: NCT01941797
Title: Experimental Peri-implant Mucositis in Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UConn Health (Other)
Collaborators: Colgate Palmolive (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: cro-2011perio-02-fp
Record Dates: First submitted 2013-09-10; First posted 2013-09-13 (Estimated); Last update posted 2017-04-26 (Actual); Status verified 2017-04

CONDITIONS: Peri-implant Mucositis; Gingivitis
MeSH Terms: conditions — Gingivitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Peri-implant mucosa (Experimental)
  Interventions: Behavioral: interruption of oral hygiene
- periodontal mucosa (Active Comparator)
  Interventions: Behavioral: interruption of oral hygiene

INTERVENTIONS:
Behavioral: interruption of oral hygiene

SUMMARY:
This is a pilot study. The investigators hypothesize that the peri-implant soft tissue response to de novo plaque accumulation is similar to that of normal gingival tissue in the same subjects.

The investigators propose to conduct a controlled clinical trial to evaluate peri-implant soft tissue response to de novo plaque accumulation in comparison to the response of gingival tissue in the same subjects

ELIGIBILITY:
Inclusion Criteria:

-Male and Female ³21 years of age.

Oral site specific inclusion criteria:

* 1) Presence of 2 implants in the maxillary or mandibular arch supporting fixed restorations in function for at least 1 year (Test)
* 2) Presence of 2 teeth in the corresponding position of the implant (Control); -3) Absence of active infections at both test and control sites
* 4) Absence of radiographic bone loss at both test and control sites
* 5) Pocket depth ≤4mm at both test and control sites
* 6) must give written informed consent.

Exclusion Criteria:

* 1) Treatment with antibiotics for any dental or medical condition within 1 month before screening
* 2) Systemic diseases that require chronic use of anti-inflammatory medications, antibiotics or anticoagulants
* 3) Ongoing medications for systemic conditions initiated <3 months before the start of the study or the requirement to take prophylactic antibiotics for invasive dental procedures
* 4) Significant organ disease including impaired kidney function, heart murmur, rheumatic fever, bleeding disorder
* 5) Active infectious diseases such as hepatitis, tuberculosis and HIV
* 6) Clinically detectable caries and periodontal disease
* 7) Tobacco use of any kind
* 8) Use of medications affecting periodontal status (diphenylhydantoin, cyclosporine etc.)
* 9) No pregnancy or lactation or expectation to become pregnant within next 3 months.

Participants will be excluded from the study or analysis if any of the following occur during the study: 1) Changes in the patient medical status or medications that met the exclusion criteria; 2) Use of antimicrobial rinses; 3) Use of irrigating devices; 4) Subject noncompliance with stent wearing during the experimental mucositis/gingivitis phase and/or Vitamin C use; 5) Use of anti-inflammatory drugs or antibiotics; 6) allergic history to common toothpaste or mouth rinse ingredients.

Acute use of acetaminophen will be permitted.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2012-09; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Gingival Crevicular fluid volume collected at baseline and weekly up to 9 weeks | 9 weeks
  The gingival crevicular fluid ( GCF) volume is assessed using Periotron unit. The GCF volume is strongly correlated with peri-implant mucosa and gingival inflammation.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Connecticut Health Center, Farmington, Connecticut, United States